CLINICAL TRIAL: NCT04946240
Title: Effects of Supervised BRACE (Balance, Resistance, Aerobic, Cognitive Exercises) Protocol on Mobility in Elderly With Fall Risk
Brief Title: Effects of Supervised (BRACE) Balance, Resistance, Aerobic &Cognitive Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00405 Umme Habiba
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Elderly Population
MeSH Terms: interventions — Braces; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised (BRACE) Group (Experimental): the self-developed protocol (BRACE) is used in the experiment with a combination of balance, resistance, aerobic and cognitive exercises for 12 weeks with repetition of different tasks
  Interventions: Other: Supervised (BRACE) Group
- Conventional Balance Exercises Group (Active Comparator): The unsupervised home plan included balance and resistance exercise was guided to conventional group
  Interventions: Other: Conventional Balance Exercises Group

INTERVENTIONS:
Other: Supervised (BRACE) Group — Supervised (BRACE) protocol include static, dynamic and anticipatory balance exercises, chair rise, stair climbing and floor transfer comes under the category of resistance exercises. 6 minutes walk test, marching in space and cycling comes in aerobic. count reverse for 50 remember 5 words, 5 animals, repeat 5 words, spell forward and backwards and cont even numbers comes in cognitive exercises.
  Arms: Supervised (BRACE) Group
Other: Conventional Balance Exercises Group — The home plan included Balance and Resistance exercises of BRACE protocol were provided to the control group but that was not supervised. Control group participants were also same assessed as the S-BRACE group. Before giving the training plan for home, it was elaborated in detail. For the convenience of participants, the BRACE protocol was also translated into Urdu and was given in the printed form. The data were collected at baseline, after 3 weeks, 6, 9 and then after 12 weeks of training
  Arms: Conventional Balance Exercises Group

SUMMARY:
In the elderly risk of fall increases due to balance dysfunction, cognitive impairment and low vision. In this research, the aim is to find the effects of Supervised BRACE (Balance, Resistance, Aerobic, Cognitive Exercises) protocol on mobility to reduce the risk of fall in the elderly. Randomized controlled trial 10-12 weeks follow-up. The sample size is 40. The subjects are divided into two groups, 20 subjects in the control group and 20 in the experimental group. The study duration is of 6 months. The sampling technique will be purposive sampling and consecutive random assignment through the sealed envelope method. Individuals of age 60-80, either gender with Berg balance score (BBS) 20-40 will be included. Individuals with musculoskeletal conditions (fractures, severe arthritis), neurological conditions like Epilepsy, Parkinson, Alzheimer's, Impaired cognition and other systemic diseases or co-morbidities will be excluded. Assessments tools that will be used in the study are Mini-Mental State Exam, Berg balance Scale, timed up and go test (TUG), elderly mobility scale, Fullerton Advanced Balance (FAB) scale, Activities of Balance Confidence.

DETAILED DESCRIPTION:
In terms of morbidity and mortality fall is a major concern in older adults. Fall is defined as unintentional contact with the ground. Tinetti in 1988 defined fall as "an event in which a person rest unintentionally on the ground or lower surface". There are many reasons for fall which can be intrinsic or extrinsic. The risk factors of fall can be ageing (e.g. cognitive impairment, poor balance or low vision), nutrition (vitamin D and calcium deficiency), medication (sedatives, antidepressants etc), environmental factors (improper shoes, poor lighting and unsafe stairs) and lack of exercise.

Previous studies considered age 60 and above in the geriatric population. The number of falls increases day by day due to balance dysfunction which is the key impairment. Age 60 and above along with any impairment or disease which makes a person weak can be included in the group of geriatric population. The fact supported by previous researches that the person who involved in rehabilitation therapies can decrease fall rate and fall associated problems. Through these rehabilitation exercises Activity of Daily Living (ADLs) can be improved and disabilities could be prevented. Wii Fit gaming system can be used to uplift lifestyle and improve balance in the geriatric population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of age 60 -80 years
* Either gender
* Berg balance score 21-40

Exclusion Criteria:

* Musculoskeletal conditions (fractures, severe arthritis grade iii and iv)
* Neurological conditions like Epilepsy, Parkinson, Alzheimer's, Impaired cognition
* Other systemic diseases or co-morbidities

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | week 12
  authentic tool to assess the balance. It is used for the assessment of static and dynamic balance. It is additionally utilized for assessment of functional balance and risk of fall in the elderly. It is a 14 Item scale, each item has a range of score from 0-4, where a high score (4) indicates a decrease in fall risk, good balance and perform task independently while a lower score (0) demonstrates poor balance, increased danger of fall and totally dependent. 56 are the highest score of berg balance
Montreal Cognitive Assessment (MoCA) | week 12
  The Montreal Cognitive Assessment (MoCA) is used for the screening of cognitive impairment. There is no effective instrument for the early detection of mild cognitive changes. MoCA is a successful screening test Scores of MoCA ranges from 0-30. Interpretation of MoCA indicates that score of 26 and above normal, 18 - 25 score indicates mild cognitive impairment, 10 - 18 score considered moderate cognitive impairment while <10 considered severe cognitive impairment exists for the screening of mild cognitive impairment.
The Timed Up and Go Test | week 12
  The Timed Up and Go Test (TUG) is a basic, reasonable and cheap method that was created to assess the mobility and gait in the elderly. The TUG involves fundamental regular movements: stand up from a seat, walking a distance of 3 meters, pivot, move back, and take a seat once again. The result is the time taken to play out this arrangement of developments.
  The interpretation of TUG demonstrates that individuals with TUG score <10 seconds are highly mobile, <20 seconds are generally independent and > 20 for mobility impairment
ACTIVITIES-SPECIFIC BALANCE CONFIDENCE | week 12
  The Activities-specific Balance Confidence (ABC) scale was produced to evaluate the confidence level in performing Score of ABC scale ranges from 0%-100%, 0% means (no confidence) and 100% means (absolutely good). The interpretation of ABC scale demonstrates >80% shows good level of confidence in physical activity, 50-80% indicates a moderate level of confidence and <50% shows a low level of confidence in physical working specific task without losing balance or getting to be unsteady.
ELDERLY MOBILITY SCALE | week 12
  The Elderly Mobility Scale (EMS) is a simple and quick tool used for the assessment of mobility and function in elderly. EMS is the 7-item scale with the total score of 20. The interpretation of EMS demonstrates , individuals with score >14 are perform their ADLs independently with good mobility, score ranges between 10-13- these individuals are at borderline according to their safe mobility and independence while score < 10 are generally dependent in performing ADLs and have poor mobility
FULLERTON ADVANCE BALANCE (FAB) SCALE | week 12
  Fullerton Advanced Balance (FAB) is a valid and reliable scale used for the assessment of balance in higher-working elderly. Both static and dynamic balance can be measured through FAB. The test was found to separate among members of fluctuating abilities of balance. FAB is 10-item scale consists of 5-point ranged (0-4) with total score of 0-40 points possible (higher scores are better). Items are scored on a 5-point ordinal scale (0-4).

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Chakwal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masud T, Morris RO. Epidemiology of falls. Age Ageing. 2001 Nov;30 Suppl 4:3-7. doi: 10.1093/ageing/30.suppl_4.3. No abstract available. PMID 11769786
- [Background] Afridi A, Malik AN, Ali S, Amjad I. Effect of balance training in older adults using Wii fit plus. J Pak Med Assoc. 2018 Mar;68(3):480-483. PMID 29540893
- [Background] Ungar A, Rafanelli M, Iacomelli I, Brunetti MA, Ceccofiglio A, Tesi F, Marchionni N. Fall prevention in the elderly. Clin Cases Miner Bone Metab. 2013 May;10(2):91-5. PMID 24133524
- [Background] Zhuang J, Huang L, Wu Y, Zhang Y. The effectiveness of a combined exercise intervention on physical fitness factors related to falls in community-dwelling older adults. Clin Interv Aging. 2014;9:131-40. doi: 10.2147/CIA.S56682. Epub 2014 Jan 10. PMID 24453483
- [Background] Heyn P, Abreu BC, Ottenbacher KJ. The effects of exercise training on elderly persons with cognitive impairment and dementia: a meta-analysis. Arch Phys Med Rehabil. 2004 Oct;85(10):1694-704. doi: 10.1016/j.apmr.2004.03.019. PMID 15468033
- [Background] Steadman J, Donaldson N, Kalra L. A randomized controlled trial of an enhanced balance training program to improve mobility and reduce falls in elderly patients. J Am Geriatr Soc. 2003 Jun;51(6):847-52. doi: 10.1046/j.1365-2389.2003.51268.x. PMID 12757574
- [Background] Muir SW, Berg K, Chesworth B, Speechley M. Use of the Berg Balance Scale for predicting multiple falls in community-dwelling elderly people: a prospective study. Phys Ther. 2008 Apr;88(4):449-59. doi: 10.2522/ptj.20070251. Epub 2008 Jan 24. PMID 18218822
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946